CLINICAL TRIAL: NCT05816304
Title: Evaluating the Effectiveness of Digital Cognitive Behavioral Therapy for Insomnia in Frontline Health Care Workers (The HCW-CBTi Study): A 2-arm, Pragmatic, Prospective, Parallel Randomized Controlled Trial
Brief Title: Effectiveness of Digital Cognitive Behavioral Therapy for Insomnia in Frontline Health Care Workers (The HCW-CBTi Study)
Acronym: HCW-CBTi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-5619
Record Dates: First submitted 2023-03-30; First posted 2023-04-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-08

CONDITIONS: Insomnia; Post Traumatic Stress Disorder; Anxiety Disorders; Depression
Keywords: Insomnia,; sleep health,; Cognitive Behavioral Therapy; Digital Cognitive Behavioral Therapy; Health Care Workers
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Two-arm, pragmatic prospective, parallel, multi-center, randomized controlled trial (RCT)
Who Masked: Participant
Masking Description: Participants will be randomized and allocated to either the intervention or attention control arm of the trial. Randomization will be centrally controlled, and allocation will be concealed using a secure, web-based randomization using the Research Electronic Data Capture (REDCap) platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Digital CBTi will be offered using the SleepioTM website and supporting Sleepio™ app (Big Health Ltd., London, UK) via 6 sessions training program (spanning 6 to 12 weeks), lasting an average of 20 minutes each, unlocked weekly. The participant will receive the Sleepio intervention as soon as they become assigned.
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy for Insomnia (dCBTi)
- Attention Control arm (No Intervention): Participants in the control group will have access to online the sleep diary and sleep education material for 12 weeks, without the CBTi intervention by the Sleepio™ app (Big Health Ltd., London, UK). They will start the digital cognitive behavioral therapy for insomnia (dCBTi) intervention 12 weeks after the initial enrollment.

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioral Therapy for Insomnia (dCBTi) — Digital CBTi is a computer-based cognitive behavioral therapy that provides strategies to improve sleep and daytime function (concentration, productivity) and decreases symptoms of sleep-related attributions, night-time thought content in individuals with insomnia. It is easily accessible with any internet-connected device, eg, computer, tabs, and smartphones.
  Other Names: Sleepio
  Arms: Intervention arm

SUMMARY:
The COVID-19 pandemic has resulted in increased workload and concerns about personal and family safety for frontline healthcare workers (HCWs), which can lead to decreased well-being and worsening mental health. Sleep disruption is particularly prevalent among HCWs providing frontline COVID-19 care. It can have direct consequences on their cognitive and emotional functioning, as well as on patient safety. Cognitive Behavioral Therapy for insomnia (CBTi) is a first-line treatment for insomnia. It has been shown to improve sleep health and wellbeing in the general population. However, there are significant barriers to delivering CBTi to frontline HCWs, including limited availability of trained sleep therapists and high costs. To address this, a Canada-wide randomized controlled trial is developed to determine the effectiveness of a digital CBTi program on the sleep health, mental health, wellness, and overall quality of life of frontline HCWs caring for COVID-19 patients. This study may provide an easily accessible and scalable sleep health intervention that can be included as part of a national and global response to the COVID-19 pandemic.

DETAILED DESCRIPTION:
Sleep disruption is prevalent in frontline healthcare workers (HCWs), of which more than 30% are physicians and nurses. The ongoing COVID-19 crisis has caused decreasing well-being and worsening mental health. Frontline HCWs involved in the management of patients with COVID-19 are nearly 3 times more likely to experience insomnia than anxiety or depression. It can have direct consequences on cognitive and emotional functioning and well-being, which impacts the safety of the patients. Insomnia is a health problem that may be appropriately treated with a less resource-intensive solution. Hypnotics can be considered for short-term use for severe insomnia but it is not free of psychological and/or physical dependence, tolerance, substance misuse, and sleepiness. Therefore, non-pharmacological sleep therapies such as CBTi may be advantageous for improving sleep health, HCW wellness, and in preventing burnout.

Cognitive Behavioral Therapy for insomnia (CBTi) is currently a first-line therapy for adults with sleep disorders including insomnia and other sleep health disruptions. The principles and specific elements of CBTi include stimulus control, sleep hygiene, relaxation therapy, cognitive re-appraisal, and sleep restriction techniques. Delivering CBTi to frontline HCWs is associated with significant barriers including the limited availability of trained sleep therapists and the high cost of receiving face-to-face treatment. Digital CBTi can be easily accessed while maintaining physical distancing, and is less resource intensive than traditional CBTi, while providing symptom self-management and ongoing coach-tailored feedback. Recently, digital CBTi (Sleepio™, Big Health Ltd., London, UK) was made available free of charge to over 1 million frontline COVID-19 HCWs in the United Kingdom's National Health Service for the duration of the COVID-19 pandemic. Indeed, CBTi has already been shown to be effective for patients with insomnia in the general population, but it has not been evaluated amongst HCWs during a pandemic. We propose a national RCT amongst frontline HCWs taking care of patients during the COVID19 era to determine the effect of a digital CBTi program (SleepioTM) on their sleep health, mental health, wellness domains, and overall HRQL.

ELIGIBILITY:
Inclusion Criteria:

* Health care workers with probable insomnia disorder, as indicated by a score of 16 or lower on the Sleep Condition Indicator (SCI),
* Self-identify as being involved in frontline management of patients;
* Access to a mobile phone or a computer with Internet access.

Exclusion Criteria:

* Participants requiring urgent CBT treatment as per their health care provider,
* Participants received CBT in the past 3 months
* Participants participating in other psychological treatments and/or drug trials during the study;
* Self-reported additional sleep related disorders: sleep apnea or restless legs syndrome;
* Significant other significant medical or psychiatric conditions e.g. life threatening (e.g. cancer), neurological conditions (e.g. epilepsy); severe depression , active suicide intent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessing changes in the nature and severity of insomnia: | 12 weeks
  Change in score on the Insomnia Severity Index (ISI ) from baseline to 12 weeks. ISI is a 7-item self-report questionnaire that assesses insomnia's nature, severity, and impact. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. The score can be classified in the following way:
  the total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "subthreshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe).

SECONDARY OUTCOMES:
Sleep Condition Indicator | 12 weeks
  It is an eight-item rating scale that was developed to screen for insomnia disorder based on DSM-5 criteria. Each item was scored on a 5-point scale (0-4), with lower scores, in the 0-2 range, reflecting putative threshold criteria for insomnia disorder. The possible total score ranges from 0 to 32, with higher values than 16 indicative of better sleep.
  The SCI is valid, reliable, and sensitive to change.
Patient Reported Outcomes Measurement Information System(PROMIS ) Sleep Disturbance | 12 weeks
  The PROMIS Sleep Disturbance is an eight-item scale that assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance. The raw scores on the 8 items should be summed to obtain a total raw score.
Patient Reported Outcomes Measurement Information System(PROMIS ) Sleep Related Impairment | 12 weeks
  The PROMIS Sleep-Related impairment is an eight-item scale that focuses on self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance. The raw scores on the 8 items should be summed to obtain a total raw score.
Generalized Anxiety Disorder (GAD) 7 | 12 weeks
  The GAD-7 is a valid and efficient tool for screening and assessing the severity of generalized anxiety disorder (GAD) in clinical practice and research. Screening for anxiety disorders, a score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder; The following cut-offs correlate with the level of anxiety severity:
  * Score 0-4: Minimal Anxiety
  * Score 5-9: Mild Anxiety
  * Score 10-14: Moderate Anxiety
  * Score greater than 15: Severe Anxiety.
Warwick Edinburgh Mental Wellbeing Scale(WEMWBS ) | 12 weeks
  14 items to measure feeling and functional aspects of mental well-being. The WEMWBS is scored by summing the scores for each of the 14 items, which are scored from 1 to 5. The 14-item scale WEMWBS has 5 response categories, summed to provide a single score. Scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.
Work And Social Adjustment Scale (WSAS) | 12 weeks
  5 items to measure functional impairment attributed to a given disorder.5 items can be scored from 0 to 8. A score of all Items will be summed up. WSAS score >20 reflects severe or worse psychopathology., 10 to 20 reflects significant functional impairment but less severe clinical symptomatology and <10 appears to signify subclinical disorders populations.
Impact of Event Scale | 12 weeks
  22 items to measure current subjective distress due to traumatic life events. The Impact of Event Scale has a scoring range of 0 to 88and a score above 24 is meaningful. A score of 24 or more will have partial PTSD or at least some of the symptoms. A score of 33 and above is a probable diagnosis of PTSD. A score of 37 or more is high enough to suppress the immune system's functioning.
Work Productivity and Activity Impairment Questionnaire | 12 weeks
  It consists of 6 items to measure impairments in works. The sum of specific health problem impairment and impairment due to other health reasons is equal to impairment due to all health reasons. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Maslach Burnout Inventory - Human Service Survey | 12 weeks
  22 items to measure burnout in medical professionals. Responses are scored on a six-point Likert scale, ranging from 0 = never to 6 = every day, for each subscale, and tabulated into three tiers (low, moderate, or high). Emotional Exhaustion (EE)-9 questions, Depersonalization (DP)-5 questions, and self-perceived lack of Personal Accomplishment (PA)-8 questions.
  Based on the reference ranges provided with the MBI-HSS: for EE, low (0-16), moderate (17-26), and high (≥27); for DP, low (0-6), moderate (7-12) and high (≥13), and finally, for PA, low (≤31), moderate (32-38) and high (≥39). Burnout was defined by the updated Maslach-recommended criteria of "high EE and high DP" or "high EE and low PA"
Patient Global Impression Scale | 12 weeks
  PGIC is a 7-point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." PGIC is commonly used to evaluate the overall improvement or change in symptoms following treatment and is an important indicator of significant change in treatments of chronic pain.
Therapy Evaluation Questionnaire | 12 weeks
  5 items can be scored from 1 to 7. The higher score signifies the greater Depth, Smoothness, and Positivity, of therapy.
Acceptability E-scale | 12 weeks
  Acceptability E-scale has strong psychometric properties and can be useful in assessing the acceptability and usability of computerized health-related programs. The score was rated on five Likert-type scale responses; 1-strongly disagree; 2disagree; 3-not sure; 4-agree; 5-strongly agree. A score of 40 or above indicates that program iss feasible for the use.
Sleep Health Disruption | 12 weeks
  Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, FRCPC, Principal Investigator — Associate Professor, Department of Anesthesiology and Pain Medicine, Toronto Western Hospital, UHN
Locations (2):
- Canada (2):
  - Toronto Western Hospital - UHN, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario